CLINICAL TRIAL: NCT06413576
Title: The Clinical Utility of Homocysteine in Critically Ill Preeclampsia Patients
Brief Title: Homocysteine in Critically Ill Preeclampsia
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R09/2024
Record Dates: First submitted 2024-04-06; First posted 2024-05-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Pre-Eclampsia; Critical Illness
MeSH Terms: conditions — Pre-Eclampsia; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- normal pregnancy: Normotensive age- matched pregnant controls
  Interventions: Diagnostic Test: homocysteine measurement
- preeclampsia: pre-eclampsia patients who are managed in ward (not critical)
  Interventions: Diagnostic Test: homocysteine measurement
- critically ill preeclampsia: pre-eclampsia patients who are admitted to intensive care unit due to severity or complications
  Interventions: Diagnostic Test: homocysteine measurement

INTERVENTIONS:
Diagnostic Test: homocysteine measurement — measuring the serum level of homocysteine

SUMMARY:
Preeclampsia is a disorder characterized by the new onset of hypertension and proteinuria typically presenting after 20 weeks of gestation. Elevated circulating homocysteine is a risk factor for endothelial dysfunction and vascular diseases such as atherosclerosis and occlusive disorders. Our study is to investigate the association between elevated blood homocysteine levels and complications in pregnant women in order to conclude the clinical utility of homocysteine as a marker of severity in the cases of pre-eclampsia.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy are an important cause of morbidity and mortality among mothers and infants. Preeclampsia is a pregnancy-related hypertensive disorder occurring usually after 20 weeks of gestation. It is associated with fetal growth restriction, low birth weight, preterm birth, respiratory distress syndrome, and admission to a neonatal intensive care unit. According to a systemic review and meta-analysis published in 2013, preeclampsia has a noticeable relationship with an increased risk of developing hypertension, ischemic heart disease, and cerebrovascular accident in later life.

There is already abundant evidence indicating that elevated serum homocysteine levels may be related to the risk of coronary, cerebral, and peripheral arterial diseases. Elevated circulating homocysteine is a risk factor of endothelial dysfunction and vascular diseases such as atherosclerosis and occlusive disorders. Normally, homocysteine levels decline throughout pregnancy and since the vascular alterations brought on by homocysteine are comparable to those brought on by hypertensive disorders of pregnancy, it can be assumed that high levels of homocysteine are linked to the hypertensive disorder spectrum. Homocysteine has been shown to produce oxidative stress and endothelial dysfunction, endothelial cell injury and thrombus formation and thereby producing pre-eclampsia.

Estimation of homocysteine may help to predict and prevent pre-eclampsia and eclampsia, thus reducing the undesired outcome of pregnancy.

Among various studies, there is a lack of consistency in the reported results that support the link between maternal homocysteine concentrations assessed throughout each of the three trimesters of pregnancy and difficulties caused by the placenta.

our study investigate the relation between the level of homocysteine and severity of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed by preeclampsia will be included in light of the following diagnostic criteria (blood pressure more than 140\90 mm\Hg on 2 occasions at least 4 hours apart after 20 weeks' gestation in a previously normotensive patient accompanied by Protein/creatinine ratio ≥0.3 .

Exclusion Criteria:

* Essential hypertension suggested by history or documentation of hypertension in pre pregnant state or hypertension before 20 weeks of gestation.
* Cardiovascular or renal failure
* Liver failure
* Diabetes mellitus
* Inflammatory or infective disorders
* History or documentation of epilepsy in prepregnant state
* Space occupying lesion in brain like tuberculoma or brain tumor
* Trauma to brain
* Hyperpyrexia
* On treatment with antifolate drugs such as methotrexate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant females
Study Population: pregnant females with pre-eclampsia and within 24 hours of delivery
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
homocysteine level | within 24 hours postoperative(post delivery)
  Quantitative measurement of the serum level of homocysteine. The measurement will be done using a commercially available sandwich enzyme linked immunosorbent assay (ELIZA) kit supplied by ( Bioassay technology laboratory) according to the manufacturer's instructions.nthe results will be expressed in ng/ml. Absorbance of standards and samples were measured at 450 nm using a microtiter plate ELISA reader .

SECONDARY OUTCOMES:
Statistical correlation analysis will be done between homocysteine levels and severity of preeclampsia | within 24 hours postoperative
  the co relation between levels of homocysteine and degree of severity of preeclampsia using spearman rank correlation co efficient

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams University, Cairo, Cairo Governorate
  - Ain shams university, Cairo, Cairo Governorate

REFERENCES:
- [Background] Salam RA, Das JK, Ali A, Bhaumik S, Lassi ZS. Diagnosis and management of preeclampsia in community settings in low and middle-income countries. J Family Med Prim Care. 2015 Oct-Dec;4(4):501-6. doi: 10.4103/2249-4863.174265. PMID 26985406
- [Background] Thakur P, Bhalerao A. High Homocysteine Levels During Pregnancy and Its Association With Placenta-Mediated Complications: A Scoping Review. Cureus. 2023 Feb 20;15(2):e35244. doi: 10.7759/cureus.35244. eCollection 2023 Feb. PMID 36968916
- [Background] Chaudhry SH, Taljaard M, MacFarlane AJ, Gaudet LM, Smith GN, Rodger M, Rennicks White R, Walker MC, Wen SW. The determinants of maternal homocysteine in pregnancy: findings from the Ottawa and Kingston Birth Cohort. Public Health Nutr. 2020 Dec;23(17):3170-3180. doi: 10.1017/S1368980019004002. Epub 2020 Mar 19. PMID 32188521
- [Background] Aubard Y, Darodes N, Cantaloube M. Hyperhomocysteinemia and pregnancy--review of our present understanding and therapeutic implications. Eur J Obstet Gynecol Reprod Biol. 2000 Dec;93(2):157-65. doi: 10.1016/s0301-2115(00)00282-7. PMID 11074137